CLINICAL TRIAL: NCT04115215
Title: Pre-FRONTal Brain STability, Key for Action Against Disability in AGing: The FRONT STAGE Project
Brief Title: Pre-FRONTal Brain STability, Key for Action Against Disability in AGing
Acronym: FRONT STAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Parc Sanitari Pere Virgili (Other)
Collaborators: Institute for Photonic Sciences - ICFO (Unknown); Hospital de la Ribera (Other); Fundacio Ictus Malaltia Vascular (Other); Institut Català de la Salut (Other); Vall d'Hebron Research Institute (sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FRONT STAGE (PI19/00734)
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Impairment; Motoric Cognitive Risk Syndrome
Keywords: Older adults; Cognitive impairment; Motoric Cognitive Risk Syndrome; Physical disfunction; Multi-component physical exercise program; Transcranial electrical stimulation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigators performing the follow-up assessments will be blind to randomization. In light of the difficulty to guarantee a complete blinding, these investigators will record if blinding is disclosed by participants during the interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Physical exercise (PE)
  Interventions: Behavioral: Physical exercise (PE)
- Arm 2 (Experimental): Transcranial current stimulation (tCS)
  Interventions: Behavioral: Physical exercise (PE); Device: Transcranial current stimulation (tCS)
- Control (Active Comparator): Educational sessions on healthy aging
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Physical exercise (PE) — This arm includes 10 sessions of multi-component exercise sessions (including aerobic, resistance, flexibility, dual-tasking) of 1 hour/week of functional group exercise, directed to foster empowerment for subsequent continuation of exercise in community-dwelling older adults referred by primary care to a geriatrician and an expert physical therapist. Participants will receive a leaflet with instructions to perform five strength-based exercises and instructors will recommend participants to perform the exercises and walk at least 15 minutes daily.
  Arms: Arm 1; Arm 2
Device: Transcranial current stimulation (tCS) — This arm includes 1 application/week for 10 weeks during PE, through an adapted commercial helmet. Transcranial current stimulation (tCS) is a neural stimulation technique based on electrical stimulation of selected parts of the brain with direct or alternated electrical current (tDCS or tACS) of very low intensity of 1,5 milliamps (mA), using one or more electrodes placed on the skull. tCS is non-invasive (no surgical procedures) and it is painless, as applied in the proposed protocols.
  Arms: Arm 2
Other: Control — Participants of similar profile, randomized to the control group, will undergo weekly 30 minutes educational sessions on healthy aging, including relevant aspects of nutrition, self-care, physical activity, plus measurement of blood pressure, heart rate and peripheral oxygen Hb saturation. These participants will be offered to join the PE program after the 6-months follow-up (end of the study).
  Arms: Control

SUMMARY:
Cognitive and mobility impairments are critical contributors to dementia and disability in older adults, and can be caused by neurodegenerative and neurovascular changes at the pre-frontal (PF) brain areas. In a previous technological project funded by ISCiii, the investigators adapted a non-invasive, point-of-care optical methods (fNRIS/fDCS technology) to study PF metabolism and blood flow activation during cognitive and motor tasks, in older adults with and without cognitive impairment. These methods are sensitive to change after physical exercise (PE) and after selectively and safely stimulating PF areas with electrical transcranial direct current stimulation (tCS). PE and tCS have shown benefits for cognition and mobility in the elderly, but their prolonged effect on PF hemodynamic activation has not been studied. Understanding the specific action of these interventions on the brain, and their clinical cognitive and motor impact, is key to fine-tune appropriate treatment strategies.

The FRONT STAGE project aims to compare, through a 3 arms single-blind randomized clinical trial, the impact of a 10 weeks, 1 hour/week program of PE (arm 1) Vs PE+tCS (arm 2) and Vs a control group (arm 3, healthy aging sessions and control of cardiovascular risk factors). The PE program is already implemented in primary care, as part of another previous project of the investigators' research group. Outcomes will include the optical measurement of PF metabolism and blood flow and clinical measures of cognitive and physical function. Front STAGE project will recruit 93 older adults with cognitive impairment and slow gait, but without dementia or disability in the activities of daily living (N=31 per arm). They will receive a comprehensive geriatric assessment at baseline, together with the optical, cognitive and physical measures, and will be follow-up at 3 and 6 months. Weekly physical activity through accelerometry will be controlled in analyses.

FRONT STAGE project centered on aging and the prevention of dementia and disability, will provide, translationally, more evidence to support and enlarge the clinical application of these interventions, and will contribute to foster further research in this field.

ELIGIBILITY:
Inclusion Criteria:

1. older adults (65 years or older)
2. with Motoric Cognitive Risk Syndrome
3. characterized by impaired cognition (which in our case will be confirmed with a Spanish version of the Montreal cognitive Assessment (MOCA), score between 26 and 21)
4. mobility impairment (measured as slow gait speed<0.8 m/s)
5. without diagnosed clinical neurological or psychiatric diseases
6. with a preserved functional status for the activities of daily living
7. who can walk without help from third parties

Exclusion Criteria:

1. a diagnosis of dementia
2. advanced/terminal disease (life expectancy<1 year)
3. contraindications to exercise and tCS
4. unwilling to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2023-03-23 (Estimated); Study Completion 2023-03-23 (Estimated)

PRIMARY OUTCOMES:
Changes in hemoglobin oxygenation during functional tasks, as measured using fNIRS+fDCS optical techniques. | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  Our primary outcome will be prefrontal hemoglobin oxygenation during a) cognitive tests, such as phonetic verbal fluency and calculations (2-forward and 3-backward counting), b) normal gait, c) dual task (walking while counting).
  All the measures will be controlled for extra-cerebral and systemic contributions due to variations in heart-rate, oxygen saturation, respiration rate and end-tidal carbondioxide. Various measures such as those derived from accelerometers to account for potential motion artifacts will be also utilized, followed by a multi-subject analysis.

SECONDARY OUTCOMES:
Cognitive executive function tests - Phonetic Verbal Fluency | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  Phonetic verbal fluency will be measured by scoring total number of words (not repeated) per unit of time, with higher rates revealing better performance.
Rey Auditory Verbal Learning Test (RAVLT) | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  Rey Auditory Verbal Learning Test (RAVLT) is a validated neuropsychological test used to assess verbal memory function.
Cognitive executive function tests - SDMT | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  The symbol-digit modalities test (SDMT) is a symbol substitution neuropsychological test that examines a person's attention and speed of processing. Higher scores will indicate better performance.
Physical function | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance), aggregated from the different subtests.
Motor function | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  "Dual task" measure: cost of gait speed reduction when a cognitive task (verbal fluency) is associated during gait, compared to gait alone.
Cognitive executive function tests - Digit span | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  The digit span is a widely used neuropsychological test to assess attention and working memory.
Cognitive executive function tests - Trail Making Test | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  Trail Making Test (TMT A and B) will be perform to assess executive function (attention).

OTHER OUTCOMES:
Spatial temporal parameters of gait | Baseline (prior to intervention), 3 and 6 months after completion of the intervention.
  Step length, width and cadence; using the portable 4 meters Protokinetics Zeno computerized carpet.
Total time of daily physical activity | 7 consecutive days (arms 2 & 3) just after the start of the intervention.
  ActivPal devices will be applied for 7 consecutive days to monitor physical activity outside and between exercise sessions, and also in the control group, in order to subsequently adjust the analyses for the activity performed out of the exercise sessions.
Clinical comorbidity | Baseline.
  The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as hospital abstracts data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
Nutritional status | Baseline.
  The Mini Nutritional Assessment Short Form (MNA®-SF) is an effective tool to help identify patients who are malnourished or at risk of malnutrition. Scores range from: 12-14 points, Normal nutritional status; 8-11 points At risk of malnutrition; 0-7 points Malnourished.
Demographics | Baseline.
  Age, gender, education, former profession, marital status, living situation and physical barriers, presence of a valid caregiver.
Self-reported quality of life | Baseline
  EuroQol-5D is a standardized instrument for measuring generic health status. It has been widely used in population health surveys, clinical studies, economic evaluation and in routine outcome measurement in the delivery of operational healthcare. This instrument is designed for self-completion and as such captures information directly from the respondent, thereby generating data that conforms with the general requirement of all Patient Reported Outcome (PRO) measures. Total score will be used, with higher scores revealing higher quality of life.
Body Mass Index | Baseline
  Weight & Height will be collected and computed to obtain Body Mass Index.
Depressive symptoms | Baseline
  The Yesavage GDS-15 items assesses depressive symptoms. The scale consists of 15 yes/no questions. Each question is scored as either 0 or 1 points. The following general cutoff may be used to qualify the severity of depressive symptoms: normal 0-4, >=5 possible depression.
Quality of sleep | Baseline
  Total score of the Jenkins questionnaire will be used to estimate quality of sleep. This questionnaire consists of 4 items rated on a 6-point scale. The 4 items ask how frequently during the previous 4 weeks the respondent experienced difficulty falling asleep, difficulty staying asleep, waking up several times per night, and waking up feeling tired and worn out after the usual amount of sleep. A dichotomous index is computed and coded as 1 if the respondents reported that any of the above sleep disturbances occurred 15 or more nights during the previous 4 weeks or as 0, if not. The selection of 15 nights as the cut-off point for sleep disturbance was based on criteria from the DSM-IV-TR, which stipulate that difficulty maintaining/initiating sleep or non-restorative sleep should be present for 3 or more nights per week for at least 1 month. A similar cut-off point for sleep disturbance was used in previous studies.
Drugs | Baseline
  Total number of drugs prescribed.
Hypertension | Baseline
  Diagnosis of hypertension (yes / no) will be collected as a cardiovascular risk factor.
Cholesterol | Baseline
  High cholesterol (yes / no) will be collected as a cardiovascular risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Inzitari, PhD, Principal Investigator — Parc Sanitari Pere Virgili - Vall d'Hebron Institute of Research
Locations (5):
- Spain (5):
  - The Institute of Photonic Sciences (ICFO), Castelldefels, Barcelona
  - Hospital Universitario La Ribera, Alzira, Valencia
  - Institut Català de la Salut, Barcelona
  - Parc Sanitari Pere Virgili, Barcelona
  - Fundació Ictus, Barcelona

IPD SHARING:
Plan to Share IPD: No